CLINICAL TRIAL: NCT06402838
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose, Multicenter, Parallel-Group Study to Investigate the Safety, Tolerability, and the Effect of RO7269162 on Amyloid and Non-Amyloid Disease-Related Biomarkers Following Daily Oral Administration in Participants at Risk for or at the Prodromal Stage of Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety and Biomarker Effects of RO7269162 in Participants at Risk for or at the Prodromal Stage of Alzheimer's Disease (AD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BP44745
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7269162 (Experimental): Participants will receive daily doses of RO7269162 for up to 72 weeks.
  Interventions: Drug: RO7269162
- Placebo (Placebo Comparator): Participants will receive daily doses of placebo for up to 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7269162 — Participants will receive daily doses (one of three dose levels) of RO7269162 for up to 72 weeks.
  Arms: RO7269162
Drug: Placebo — Participants will receive daily doses of placebo for up to 72 weeks.
  Arms: Placebo

SUMMARY:
This clinical trial is recruiting people who either are at risk of AD - have build-up of beta-amyloid, but have no clinical symptoms, or with a diagnosis of mild cognitive impairment. People can take part if they have a certain level of plaques (beta-amyloid) in the brain, shown by a positron emission tomography (PET) scan, a medical imaging technique in which tracers are injected to visualize specific pathological processes in the brain. People who take part in this clinical trial (participants) will be given RO7269162 OR placebo for up to about 1 and a half years. The clinical trial team will see them every 3 weeks in the first 3 months and then every 6 weeks until the end of the trial. These hospital visits will include checks to see how the participant responds to the treatment and any side effects they may have. The total time of participation in the clinical trial will be 90 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18 to 35 kg/m^2 inclusive at screening
* Participants must be either cognitively unimpaired or with a diagnosis of MCI due to AD, according to the National Institute on Aging - Alzheimer's Association (NIA - AA) research framework
* Clinical Dementia Rating-Global Score (CDR-GS) of 0 or 0.5
* Positive amyloid PET scan based on a cut-off of ≥24 CL units
* Availability of a person (referred as a "study partner" throughout the protocol) who: (a) has frequent and sufficient contact (e.g., minimum twice a week in-person, via telephone, video calls, by e-mail or other electronic means) with the participant, and is willing and able to provide accurate information regarding the participant's cognitive and functional abilities, signs the necessary ICF(s), and has sufficient cognitive capacity to accurately report on the participant's cognitive and functional abilities; (b) is in sufficient good general health to have a high likelihood of maintaining the same level of interaction with the participant and participation in study procedures throughout the duration of the study; and (c) is fluent in the language of the tests used at the study site. Please note that the study partner does not need to be a family member. Every effort should be made to keep the same study partner throughout the study
* In case of treatment with symptomatic AD medications, dosing regimen must be stable for at least eight weeks prior to baseline

Exclusion Criteria:

* Any medical history or evidence of a condition other than AD that may affect cognition
* History or presence of significant cardiovascular conditions and/or significant hematological disease
* History or presence of chronic kidney disease and/or impaired hepatic function
* Uncontrolled/poorly controlled diabetes
* History of or active inflammatory bowel disease
* Have received any passive or active immunotherapy (immunoglobulin) or other long-acting biologic agent that is under evaluation or approved to prevent or postpone cognitive decline administered within 1 year prior to baseline, and/or any other investigational treatment within five half-lives or 16 weeks prior to screening, whichever is longer

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | up to week 72
Change from baseline in brain amyloid load, as measured by amyloid positron emission tomography ( PET) scan | Baseline to Week 72

SECONDARY OUTCOMES:
Change from baseline in Aβ37 in cerebrospinal fluid (CSF) | Baseline to Week 72
Change from baseline in Aβ38 in CSF | Baseline to Week 72
Change from baseline in Aβ40 in CSF | Baseline to Week 72
Change from baseline in Aβ42 in CSF | Baseline to Week 72
Change from baseline in Aβ40 in plasma | Baseline to Week 72
Change from baseline in Aβ42 in plasma | Baseline to Week 72
Plasma concentrations of RO7269162 | Baseline to Week 72
CSF concentrations of RO7269162 | Baseline to Week 72

OTHER OUTCOMES:
Change from baseline in p-tau 217 in plasma | Baseline to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (48):
- Chile (2):
  - Centro de Investigación Clínica UC-CICUC, Santiago
  - Hospital Clinico Univ de Chile, Santiago
- Denmark (2):
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, Koebenhavn Oe
- France (8):
  - Groupement Hospitalier Est - Hôpital Neurologique, Bron
  - Hopital B Roger Salengro, Lille
  - Hôpital de la Timone, Marseille
  - Hôpital Lariboisière, Paris
  - CHU de Rouen Hopital, Rouen
  - Hop Guillaume Et Rene Laennec, Saint-Herblain
  - Hôpital Robertsau, Strasbourg
  - Gerontopole, Toulouse
- Germany (3):
  - Ambulates Gesundheitszentrum der Charité GmbH, Berlin
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - TUM Klinikum rechts der Isar;Ambulanz für neurokognitive Erkrankungen, München
- Italy (4):
  - Ospedale Cardinale Panico, Tricase (LE), Apulia
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fondazione Istituto Neurologico Mondino IRCCS, Pavia, Lombardy
- Poland (9):
  - ProNeuro Centrum Medyczne, ?ory
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - NZOZ Vitamed, Bydgoszcz
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - EUROMEDIS Sp z o o, Szczecin
  - ETG Neuroscience Sp. z o.o., Warsaw
  - NZOZ WCA, Wroc?aw
- South Korea (2):
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
- Spain (11):
  - Hospital General De Catalunya, Sant Cugat del Vallès, Barcelona
  - Policlínica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamaca, Salamanca
  - Fundacio ACE, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Victoria Eugenia, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario la Fe, Valencia
- United Kingdom (7):
  - Re:Cognition Health Birmingham, Birmingham
  - Surrey and Borders NHS Foundation Trust, Chertsey
  - Scottish Brain Sciences, Edinburgh
  - RE:Cognition Health, London
  - Charing Cross Hospital, London
  - Manchester Mental Health and Social Care Trust, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing